CLINICAL TRIAL: NCT05456152
Title: National, Multicenter, Open, Single-arm, Phase III Clinical Trial to Evaluate the Safety and Efficacy of Zolpidem in the Long-Term Treatment of Insomnia.
Brief Title: Safety and Efficacy of Zolpidem in the Long-Term Treatment of Insomnia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMS0222- SERENA
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Chronic Insomnia
Keywords: Chronic insomnia; Sleep disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — Administration, Sublingual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sublingual zolpidem (Experimental): 1 sublingual tablet (5mg) 30 minutes before bed time during 60 days.
  Interventions: Drug: Sublingual Tablet

INTERVENTIONS:
Drug: Sublingual Tablet — Sublingual zolpidem - 1 sublingual tablet 30 minutes before bed time.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of sublingual zolpidem during the long-term treatment of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Age between 18 to 64 years;
* Participants diagnosed with chronic insomnia defined by difficulty in initiating or maintaining sleep in the last 3 months for at least 3 nights a week according to DSM-V criteria and confirmed by polysomnography;
* Participants with difficulty in initiating or maintaining sleep parameters.

Exclusion Criteria:

* Participants with clinical or laboratory diagnose of non-treated hypothyroidism or hyperthyroidism, kidney or liver failure;
* Known hypersensitivity to any of the formula compounds;
* Participants with other sleep disorders according to the International Classification Sleep Disorders (3rd edition), example: sleep-relate breathing disorders, circadian rhythm sleep-wake disorders, parasomnias (including history of sleep-walking after hypnotic use) and sleep related movement disorders;
* Participants using sedatives or hypnotic medications;
* Participants with current diagnosis of depression or anxiety according to the Diagnostic and Statistical Manual of Mental Disorders;
* Participants with history of drug and alcohol abuse in the past 2 years;
* Participants with current smoking habits during the night period;
* Participants who treated insomnia in the last 3 months;
* Participants who are pregnant, breastfeeding or planning to get pregnant or female participants with the potential to become pregnant who are not using a reliable method of contraception;
* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Participants with current or medical history of cancer in the last 5 years;
* Participants who participated in other research protocol in the last 12 months, unless the investigator judges that there may be a direct benefit to it.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 358 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
To assess the safety profile of sublingual zolpidem during the long-term insomnia treatment. | 60 days.
  The safety profile will be assessed considering the number and percentage of each adverse event.

SECONDARY OUTCOMES:
To evaluate daytime sleepiness in the next morning. | 60 days.
  The daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS). The scale has a score from 0 to 24 and a score more than 10 is considered as excessive daytime sleepiness.
To assess the adverse events during 7 days after the last dose administration. | 7 days.
  The safety profile will be assessed considering the number and percentage of each adverse event occurred 7 days after the last dose administration.
To assess the number of adverse events in different periods of the clinical trial. | 60 days.
  The safety profile will be assessed considering the number of adverse events during the first 30 days and from 31 to 60 days of treatment.
To assess the number of participants with adverse events in different periods of the clinical trial. | 60 days.
  The safety profile will be assessed considering the number of adverse events during the first 30 days and from 31 to 60 days of treatment.

OTHER OUTCOMES:
To assess the efficacy of sublingual zolpidem in the sleep induction. | 60 days.
  The efficacy will be evaluated considering any change in the Latency to Persistent Sleep parameter (LPS) after 60 days of treatment in comparison to the baseline measure.
To assess the efficacy of sublingual zolpidem in the improvement of sleep quality. | 60 days.
  The efficacy will be evaluated considering any change in the Sleep Efficiency parameter (SE) after 60 days of treatment in comparison to the baseline measure.
To assess the efficacy of sublingual zolpidem in the improvement of time awake before onset. | 60 days.
  The efficacy will be evaluated considering any change in the Wake After Sleep Onset parameter (WASO) after 60 days of treatment in comparison to the baseline measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No